CLINICAL TRIAL: NCT02110134
Title: A Study of the RevLite Laser System for the Treatment of Refractory Mixed Type Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN13-REV-TOP-MEL-AK
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Revlite Laser System with Topical (Experimental): Revlite Laser System for the Treatment of Melasma and hydroquinone skin care regimen
  Interventions: Device: Revlite Laser System with hydroquinone skin care regimen
- Topical (Active Comparator): Hydroquinone skin care regimen
  Interventions: Other: Hydroquinone skin care regimen

INTERVENTIONS:
Device: Revlite Laser System with hydroquinone skin care regimen — Revlite Laser System with hydroquinone skin care regimen for the Treatment of Melasma
  Arms: Revlite Laser System with Topical
Other: Hydroquinone skin care regimen — Hydroquinone skin care regimen for the Treatment of Melasma
  Arms: Topical

SUMMARY:
The purpose of this study is to compare a hydroquinone skin care regimen alone to a combination of Revlite Laser treatment with a hydroquinone skin care regimen for the treatment of melasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Fitzpatrick Skin Type III-VI
* Subjects with mixed (epidermal and dermal) type melasma diagnosed by Wood's Lamp.
* Subjects who are over the age of 18 years of age
* The subject is willing and able to comply with study instructions and return to the clinic for required visits.
* The subject's melasma has persisted for greater than 6 months

Exclusion Criteria:

* The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
* The subject has a history of cutaneous photosensitization, porphyria, and hypersensitivity to porphyrins or photodermatosis.
* The subject has any skin pathology or condition that could interfere with the evaluation or requires the use of interfering topical or systemic therapy.
* The subject has an uncorrected coagulation defect or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy).
* The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 30 days prior to entering this study.
* The subject has used photosensitizing drugs (e.g., Declomycin, sulfa antibiotics, phenothiazines, etc.) within a timeframe where photosensitization from these drugs may still be present.
* The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
* The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
* The subject has Diabetes Type 1 or 2.
* The subject has a sensitivity to hydroquinone or Retin-A.
* The subject has evidence of a compromised immune system or hepatitis.
* Has had microdermabrasion in past 3 months, other laser or Intense Pulsed Light treatment or chemical peels to the face in past 6 months, injectable fillers, topical retinoids, over-the-counter anti-aging products past 2 weeks.
* Has a history of keloids or hypertrophic scarring
* Has permanent make-up and/or is unwilling to refrain from using semi-permanent cosmetics during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rates of Adverse Events Among Patients | From study baseline to completion, approximately 1 year. However, adverse events not resolved by then will be followed up with until they are resolved.
  Adverse events were collected and reported to test the safety and efficacy of the device.

SECONDARY OUTCOMES:
Satisfaction Questionnaire | 1 month post last treatment
  Physician and subject satisfaction will be ranked on a scale from 1 to 5, where 1 is extremely dissatisfied and 6 is extremely satisfied.
Photographic Evaluation using the Global Aesthetic Improvement Scale | 1 month post last treatment
  Photos will be a taken at baseline and post treatment and then improvement assessed using the Global Aesthetic Improvement Scale. This scale ranges from 0 to 3, where 0 is 0-25% clearance from baseline photograph, 1 is 25-50% clearance from baseline photograph, 2 is 50-75% clearance from baseline photograph, and 3 is 75-100% clearance from baseline photograph.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- NY Laser and Skin Care, New York, New York, United States